CLINICAL TRIAL: NCT03503422
Title: Optimizing Chronic Low Back Pain Exercise Therapies With Cerebral Electrical Stimulation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Collaborators: Foundation for Research Support of the State of Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and low back exercise
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain, Recurrent; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (anodal) + therapeutic exercises (Experimental): Real transcranial direct current stimulation associated with therapeutic exercises
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Procedure: Real transcranial direct current stimulation + therapeutic exercises for back pain
- tDCS (sham) + therapeutic exercises (Sham Comparator): Sham transcranial direct current stimulation associated with therapeutic exercises
  tDCS: 20 minutes (30 seconds ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Procedure: Sham transcranial direct current stimulation + therapeutic exercises for back pain

INTERVENTIONS:
Procedure: Real transcranial direct current stimulation + therapeutic exercises for back pain — Real transcranial direct current stimulation associated with therapeutic exercises for back pain
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively.
  Arms: tDCS (anodal) + therapeutic exercises
Procedure: Sham transcranial direct current stimulation + therapeutic exercises for back pain — Sham transcranial direct current stimulation associated with therapeutic exercises for back pain.
  tDCS: 20 minutes (30 seconds ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion). Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively
  Arms: tDCS (sham) + therapeutic exercises

SUMMARY:
Chronic low back (CLBP) pain is an important public health and socioeconomic problem worldwide and, despite the volume of research in the area, it remains a difficult condition to treat. The Neuromatrix pain model and new findings on the pain chronification process point to a greater efficacy of treatments that address central and peripheral rather than only peripheral structures.

Transcranial direct current (tDCS) stimulation is a noninvasive neuromodulation technique that has been presenting recent advances in the treatment of chronic pain. However, when applied alone the magnitude of its effect is small in chronic musculoskeletal conditions such as chronic non-specific back pain. One option that could optimize the analgesic effect of tDCS would be the combination with therapeutic exercises, which play a central role in spinal rehabilitation programs as well as higher levels of evidence. The combination of these treatments (tDCS and exercise) may present an analgesic effect superior to the isolated interventions.

This study aims to investigate the efficacy of tDCS combined with therapeutic exercises in people CLBP for pain relief, affective aspect of pain, disability, kinesiophobia and global perception. Sixty patients will be randomized into two distinct groups to receive either tDCS (anodal) + therapeutic exercises or tDCS (sham) + therapeutic exercises for 12 sessions over a four-week period. The primary clinical outcome (pain relief) and secondary outcomes (disability, affective aspect of pain, kinesiophobia, and perception of overall effect) will be collected before treatment and four weeks, three months and six months post randomization. The data will be collected by a blind examiner to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

Complaining of back pain for more than three months. Presence of a chronic pain measurable with the number rating scale (NRS 0-10) not less than 4 during a 1 week daily NRS monitoring.

Seeking care for low back pain. -

Exclusion Criteria:

Previous surgery on the spine, spondylolisthesis Previous treatment with TENS <6 months Previous treatment with tDCS Disc herniation with nerve compression Neurological, psychiatric and rheumatologic diseases Impaired sensibility Use of pacemakers or other implanted devices Pregnancy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Four weeks after randomization
  Pain intensity will be evaluated by numerical rating scale (0-10).

SECONDARY OUTCOMES:
Quality of pain | 4 weeks, 3 and 6 months after randomization
  The Short form of the McGill pain questionnaire (SF-MPQ) consists of 15 representative words from the sensory and affective categories of the standard long form. The 6 point intensity scale and a VAS are included to provide indices of overall pain intensity.
Disability | 4 weeks, 3 and 6 months after randomization
  The Roland Morris disability questionnaire (RMDQ) is composed of 24 yes or no questions designed to assess disability related to back pain.
Tampa Scale for Kinesiophobia | 4 weeks, 3 and 6 months after randomization
  Irrational, and debilitating fear of movement and activity resulting from a feeling of vulnerability to painful injury or re-injury. Its a 17-item scale.
Global perceived effect (GPE) | 4 weeks, 3 and 6 months after randomization
  Global perceived effect is an 11 point scale that ranges from 5 (vastly worse) through 0 (no change) to 5 (completely recovered). For all measures of global perceived effect (at baseline and all follow-ups), participants were asked compared to when this episode ﬁrst started, how would you describe your back these days. A higher score indicates higher recovery from the condition.

OTHER OUTCOMES:
Anxiety | 4 weeks, 3 and 6 months after randomization
  Visual analogue scale (VAS)for anxiety assesses anxiety symptoms that we tracked as possible confounding factor.
  The VAS for general anxiety is assessed by a horizontal 100-mm-long line. The extreme left end points to no anxiety, and the extreme right end to the worst anxiety possible.
Depression | 4 weeks, 3 and 6 months after randomization
  Beck depression inventory (BDI) for depressive symptoms that we tracked as possible confounding factor.
  The BDI is a tool of self-assessment of de- pression using a questionnaire with 21 items whose in- tensity varies from 0 to 3 (higher scores indicating more depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Fuad A Hazime, PhD, Principal Investigator — Federal University of Piaui
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cavalcante PGL, Baptista AF, Cardoso VS, Filgueiras MC, Hasue RH, Joao SMA, Hazime FA. Transcranial Direct Current Stimulation Combined With Therapeutic Exercise in Chronic Low Back Pain: Protocol of a Randomized Controlled Trial. Phys Ther. 2020 Aug 31;100(9):1595-1602. doi: 10.1093/ptj/pzaa105. PMID 32526017